CLINICAL TRIAL: NCT04093570
Title: An Open-Label, Multicenter, Extension Study for Subjects Who Participated in Prior Clinical Studies of ASTX727 (Standard Dose)
Brief Title: A Study for Participants Who Participated in Prior Clinical Studies of ASTX727 (Standard Dose)
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ASTX727-06; 2024-516293-29-01 (EU CTIS Number); 2018-003942-18 (EudraCT Number)
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia; Myelodysplastic Syndromes
Keywords: cedazuridine; decitabine; MDS; CMML; AML; myelodysplastic syndromes; chronic myelomonocytic leukemia; acute myeloid leukemia; ASTX727; INQOVI
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — decitabine and cedazuridine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Main Extension Study: ASTX727 (Experimental): The recommended starting dose is the fixed-dose combination (FDC) standard dose (SD) tablet, containing 100 mg cedazuridine and 35 mg decitabine, once daily, Days 1 through 5 in 28-day cycles. Participants should receive ASTX727 at the same dose they received in the last cycle of their parent study; if an adjustment from that dose is required, a different total cycle dose may be employed, as guided by the dose adjustment guidelines in the parent study protocol.
  Interventions: Drug: ASTX727
- Substudy Arm A: ASTX727 With High-Calorie/High-Fat Breakfast Meal on Day 4 (Experimental): Participants received ASTX727 once daily on Days 1 through 5 in a 28-day cycle (Cycle 1). Participants fasted for at least 2 hours before and 2 hours after dosing on Days 1, 3, 5 and for at least 10 hours before and 4 hours after dosing on Day 2. Participants received a high-calorie/high-fat breakfast meal after an overnight fast of at least 10 hours before dosing on Day 4 and continued to fast for at least 4 hours post-dose.
  Participants continued treatment with ASTX727 in Cycle 2 onwards in the ASTX727-06 study at the Investigator's discretion, where they continued to receive ASTX727 unless there was occurrence of disease progression requiring alternative therapy, unacceptable toxicity, noncompliance, a decision to discontinue treatment, or if the participant withdraws from the study.
  Interventions: Drug: ASTX727
- Substudy Arm B: ASTX727 With Low-Calorie/Low-Fat Breakfast Meal on Day 4 (Experimental): Participants received ASTX727 once daily on Days 1 through 5 in a 28-day cycle (Cycle 1). Participants fasted for at least 2 hours before and 2 hours after dosing on Days 1, 3, 5 and for at least 10 hours before and 4 hours after dosing on Day 2. Participants received low-calorie/low-fat breakfast meal after an overnight fast of at least 10 hours before dosing on Day 4 and will continue to fast for at least 4 hours post-dose.
  Participants continued treatment with ASTX727 in Cycle 2 onwards in the ASTX727-06 study at the Investigator's discretion, where they continued to receive ASTX727 unless there was occurrence of disease progression requiring alternative therapy, unacceptable toxicity, noncompliance, a decision to discontinue treatment, or if the participant withdraws from the study.
  Interventions: Drug: ASTX727

INTERVENTIONS:
Drug: ASTX727 — ASTX727 film-coated, immediate-release FDC tablets
  Other Names: cedazuridine + decitabine; INQOVI; DEC-C

SUMMARY:
Extension study to provide ongoing long-term treatment with ASTX727 for participants who were benefitting from ASTX727 treatment in a previous Taiho (formerly Astex)-sponsored clinical study of ASTX727 (including, but not limited to ASTX727-01 [NCT02103478], ASTX727-02 [NCT03306264], ASTX727-04 [NCT03813186]), ASTX727-06 [NCT04093570] food effect substudy, ASTX727-17 [NCT04953897], and ASTX727-18 [NCT04953910] to obtain long-term safety information.

The purpose of the Food Effect Substudy was to evaluate the pharmacokinetics (PK) and safety of decitabine and cedazuridine when ASTX727 was given under fed (high-calorie/high-fat meal or low-calorie/low-fat meal) versus fasted conditions. Food Effect Substudy has now completed.

DETAILED DESCRIPTION:
Main Extension Study: Participants will attend clinic visits on Day 1 of each 28-day cycle to undergo study procedures and to be given ASTX727 tablets for Days 1-5 of that dose cycle. Participants should continue to receive the same ASTX727 dose and regimen they were receiving in the last cycle of the parent study in which they were originally enrolled. Subsequent treatment delays and/or dose reductions are at the discretion of the investigator as guided by the dose adjustment guidelines of the parent study protocol.

Food Effect Substudy: Participants received ASTX727 once daily on Days 1 through 5 followed by a 23-day treatment-free period in a 28-day cycle (Cycle 1). Participants received either a high-calorie, high-fat breakfast meal (Arm A) or a low-calorie/low-fat breakfast meal (Arm B) predose on Day 4. Participants in Arms A and B received ASTX727 on Days 1, 2, 3, and 5 in the fasted condition. Participants may continue treatment with ASTX727 in Cycle 2 onwards in the ASTX727-06 study at the Investigator's discretion, where they continued to receive ASTX727. This substudy consists of a 21-day Screening Period, a 1-cycle (28 days) Treatment Period, and a 30-day (+7 days) Safety Follow-up Period (only if the participant discontinues from the ASTX727-06 food effect substudy and does not continue to receive ASTX727 in the ASTX727-06 study).

ELIGIBILITY:
Inclusion Criteria for the Main Extension Study:

Participants must fulfill all of the following inclusion criteria:

1. Previous participation in a Taiho (formerly Astex)-sponsored ASTX727 clinical trial (including, but not limited to studies ASTX727-01, ASTX727-02, and ASTX727-04, , ASTX727-17, and ASTX727-18, and the food effect substudy of ASTX727-06) in which the participant was treated with ASTX727 and was still on active treatment with ASTX727 at the time of study completion as determined by Taiho.
2. Participant is considered to be benefitting from ASTX727 treatment in the opinion of the treating investigator at the time of parent study completion (Participants must not be withdrawn from the parent study until eligibility for this study is confirmed).
3. Participant is able to understand and comply with the study procedures and understands the risks involved in the study.
4. Participant provides legally effective informed consent before undergoing any study-specific procedure.
5. Women of childbearing potential must not be pregnant or breastfeeding and must have a negative pregnancy test at screening. Women of childbearing potential must agree to practice 1 highly effective contraceptive methods of birth control during the study and for 6 months after the last dose of study treatment, agree not to donate eggs for the purpose of reproduction during this period and must agree not to become pregnant for 6 months after completing treatment; men with female partners of childbearing potential must agree to practice 2 highly effective contraceptive measures and must agree not to father a child while receiving ASTX727 and for at least 3 months after completing ASTX727 treatment.

Inclusion Criteria for the Food Effect Substudy:

1. Participants must have a confirmed diagnosis of-

   i. Myelodysplastic syndromes (MDS) including all French-American-British subtypes (refractory anemia, refractory anemia with ringed sideroblasts, refractory anemia with excess blasts, refractory anemia with excess blasts in transformation, chronic myelomonocytic leukemia [CMML])), and participants with MDS International Prognostic Scoring System (IPSS) int-1, int-2, or high-risk MD.

   ii. Acute myeloid leukemia (AML), as diagnosed according to the 2016 World Health Organization (WHO) guidelines on acute leukemia, of any subtype except M3 (acute promyelocytic leukemia), who are not candidates for intensive chemotherapy, including participants receiving hypomethylating agent (HMA) treatment, who have a confirmed diagnosis and a prior confirmatory bone marrow report. Participants who are currently receiving HMA treatment must complete the ongoing (at the time of Screening) treatment cycle before enrolling in this study; timing of start of treatment cycle with ASTX727 is at the principal investigator's discretion.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
3. Adequate organ function defined as follows:

   1. Hepatic: Total bilirubin ≤1.5 × upper limit of normal (ULN); aspartate aminotransferase/serum glutamic-oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase/serum glutamic-pyruvic transaminase (ALT/SGPT) ≤5 × ULN.
   2. Renal: Calculated creatinine clearance ≥60 mL/min.

Exclusion Criterion for the Main Extension Study:

1. Any participant who, in the opinion of the investigator, may have other conditions, organ dysfunction, or for whom safety data from parent study participation suggests the risks of continuing treatment with ASTX727 may outweigh the benefits.

Exclusion Criteria for the Food Effect Substudy:

1. Participants with known or suspected hypersensitivity to decitabine, cedazuridine, or any of the excipients in the ASTX727 tablets.
2. Poor medical risk because of other conditions such as uncontrolled systemic diseases or active uncontrolled infections.
3. Life-threatening illness, medical condition or organ system dysfunction, or other reasons including laboratory abnormalities, which, in the Investigator's opinion, could compromise the participant's safety, interfere with the absorption or metabolism of decitabine + cedazuridine or compromise the integrity of the study outcomes.
4. Prior gastric surgery for ulcer disease, weight loss, etc, that would impair normal motility or absorption.
5. Second malignancy currently requiring active chemotherapy. To clarify, participants with breast or prostate cancer stable on or responding to endocrine therapy, are eligible.
6. Known history of human immunodeficiency virus or known seropositive for hepatitis C virus or hepatitis B virus.
7. Active uncontrolled gastric or duodenal ulcer.
8. Participants with acute promyelocytic leukemia.
9. Prior cytotoxic chemotherapy for AML except for hydroxyurea to control high white blood cell (WBC) counts.
10. Treated with any investigational drug or therapy within 2 weeks of study treatment, or 5 half-lives, whichever is longer, before the protocol-defined first dose of study treatment, or ongoing clinically significant AEs from previous treatment with investigational drug or therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Main Extension Study: Safety: Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | From date of transition into this extension study until 30 days following the last dose, up to approximately 2 years
  An adverse event (AE) is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including a clinically significant abnormal finding in laboratory tests or other diagnostic procedures), symptom, or disease temporally associated with the use of a drug, without any judgment about causality. TEAEs are defined as events that first occur or worsen on or after the date of the first study treatment until 30 days after the last dose of study treatment, or the start of an alternative anticancer treatment, whichever first.
Food Effect Substudy: AUC0-last: Area Under the Plasma Concentration-time Curve From Time Zero to Last Concentration Measured of Decitabine in the Fasted and Fed State | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours post dose on Days 2 (fasted state) and 4 (fed state) in Cycle 1 ( up to 28 days)
Food Effect Substudy: AUC0-last: Area Under the Plasma Concentration-time Curve From Time Zero to Last Concentration Measured of Cedazuridine in the Fasted and Fed State | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours post dose on Days 2 (fasted state) and 4 (fed state) in Cycle 1 (up to 28 days)
Food Effect Substudy: AUC0-last: Area Under the Plasma Concentration-time Curve From Time Zero to Last Concentration Measured of Cedazuridine-epimer in the Fasted and Fed State | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours post dose on Days 2 (fasted state) and 4 (fed state) in Cycle 1 (up to 28 days)
Food Effect Substudy: AUC0-8h: Area Under the Concentration-time Curve From Time Zero to 8 Hours of Decitabine in the Fasted and Fed State | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post dose on Days 2 (fasted state) and 4 (fed state) in Cycle 1 (up to 28 days)
Food Effect Substudy: AUC0-8h: Area Under the Concentration-time Curve From Time Zero to 8 Hours of Cedazuridine in the Fasted and Fed State | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post dose on Days 2 (fasted state) and 4 (fed state) in Cycle 1 (up to 28 days)
Food Effect Substudy: AUC0-8h: Area Under the Concentration-time Curve From Time Zero to 8 Hours of Cedazuridine-epimer in the Fasted and Fed State | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post dose on Days 2 (fasted state) and 4 (fed state) in Cycle 1 (up to 28 days)
Food Effect Substudy: AUC0-24h: Area Under the Concentration-time Curve From Time Zero to 24 Hours of Decitabine in the Fasted and Fed State | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours post dose on Days 2 (fasted state) and 4 (fed state) in Cycle 1 (up to 28 days)
Food Effect Substudy: AUC0-24h: Area Under the Concentration-time Curve From Time Zero to 24 Hours of Cedazuridine in the Fasted and Fed State | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours post dose on Days 2 (fasted state) and 4 (fed state) in Cycle 1 (up to 28 days)
Food Effect Substudy: AUC0-24h: Area Under the Concentration-time Curve From Time Zero to 24 Hours of Cedazuridine-epimer in the Fasted and Fed State | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours post dose on Days 2 (fasted state) and 4 (fed state) in Cycle 1 (up to 28 days)
Food Effect Substudy: AUC 0-inf: Area Under the Concentration-time Curve From Time Zero to Infinity of Decitabine in the Fasted and Fed State | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours post dose on Days 2 (fasted state) and 4 (fed state) in Cycle 1 (up to 28 days)
Food Effect Substudy: AUC 0-inf: Area Under the Concentration-time Curve From Time Zero to Infinity of Cedazuridine in the Fasted and Fed State | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours post dose on Days 2 (fasted state) and 4 (fed state) in Cycle 1 (up to 28 days)
Food Effect Substudy: AUC 0-inf: Area Under the Concentration-time Curve From Time Zero to Infinity of Cedazuridine-epimer in the Fasted and Fed State | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours post dose on Days 2 (fasted state) and 4 (fed state) in Cycle 1 (up to 28 days)
Food Effect Substudy: Cmax: Maximum Observed Plasma Concentration of Decitabine in the Fasted and Fed State | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours post dose on Days 2 (fasted state) and 4 (fed state) in Cycle 1 (up to 28 days)
Food Effect Substudy: Cmax: Maximum Observed Plasma Concentration of Cedazuridine in the Fasted and Fed State | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours post dose on Days 2 (fasted state) and 4 (fed state) in Cycle 1 (up to 28 days)
Food Effect Substudy: Cmax: Maximum Observed Plasma Concentration of Cedazuridine-epimer in the Fasted and Fed State | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours post dose on Days 2 (fasted state) and 4 (fed state) in Cycle 1 (up to 28 days)
Food Effect Substudy: Tmax: Time of First Occurrence of Cmax of Decitabine in the Fasted and Fed State | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours post dose on Days 2 (fasted state) and 4 (fed state) in Cycle 1 (up to 28 days)
Food Effect Substudy: Tmax: Time of First Occurrence of Cmax of Cedazuridine in the Fasted and Fed State | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours post dose on Days 2 (fasted state) and 4 (fed state) in Cycle 1 (up to 28 days)
Food Effect Substudy: Tmax: Time of First Occurrence of Cmax of Cedazuridine-epimer in the Fasted and Fed State | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours post dose on Days 2 (fasted state) and 4 (fed state) in Cycle 1 (up to 28 days)
Food Effect Substudy: T1/2: Terminal Half Life of Decitabine in the Fasted and Fed State | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours post dose on Days 2 (fasted state) and 4 (fed state) in Cycle 1 (up to 28 days)
Food Effect Substudy: T1/2: Terminal Half Life of Cedazuridine in the Fasted and Fed State | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours post dose on Days 2 (fasted state) and 4 (fed state) in Cycle 1 (up to 28 days)
Food Effect Substudy: T1/2: Terminal Half Life of Cedazuridine-epimer in the Fasted and Fed State | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours post dose on Days 2 (fasted state) and 4 (fed state) in Cycle 1 (up to 28 days)

SECONDARY OUTCOMES:
Food Effect Substudy: Percentage of Participants with Treatment Emergent Adverse Events (TEAEs), by Severity | From first dose of study drug up to 30 days after the last dose (Up to approximately 65 days)
  An AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including a clinically significant abnormal finding in laboratory tests or other diagnostic procedures), symptom, or disease temporally associated with the use of a drug, without any judgment about causality. TEAEs are defined as events that first occur or worsen on or after the date of the first study treatment (Cycle 1 Day 1) until 30 days after the last dose of study treatment, or the start of an alternative anticancer treatment, whichever first. Severity of TEAEs were graded using Common Terminology Criteria for Adverse Events Version 4.03 (CTCAE v4.03).
Food Effect Substudy: Percentage of Participants with Clinically Significant Abnormal Laboratory Values | From Day 1 up to Day 28 in Cycle 1 (Up to 28 days)
  The laboratory parameters of hematology, serum chemistry, and urinalysis were assessed.

CONTACTS AND LOCATIONS:
Locations (48):
- United States (21):
  - Compassionate Care Research Group, Fountain Valley, California
  - Boca Raton Clinical Research, Plantation, Florida
  - The University of Chicago Medical Center, Chicago, Illinois
  - The Sidney Kimmel Comprehensive Cancer Center at John Hopkins, Baltimore, Maryland
  - Cancer and Hematology Centers for Western Michigan, Grand Rapids, Michigan
  - Mayo - Rochester, Rochester, Minnesota
  - Hackensack Medical Center - 06 FE Study, Hackensack, New Jersey
  - Hackensack Medical Center, Hackensack, New Jersey
  - Rosewell Park Cancer Institute, Buffalo, New York
  - Roswell Park Cancer Institute - 06 FE Study, Buffalo, New York
  - Gabrail Cancer Center Research - 06 FE Study, Canton, Ohio
  - Gabrail Cancer Center Research, Canton, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Charleston Hematology Oncology Associates, Charleston, South Carolina
  - Vanderbilt - Ingram Cancer Center, Nashville, Tennessee
  - Baylor Scott White University Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - May Cancer Center, San Antonio, Texas
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Seattle Cancer Care Alliance/Fred Hutchinson Cancer Research Center, Seattle, Washington
- Armenia (4):
  - Erebuni Medical Center, Yerevan
  - Hematology Center After Prof. R. Yeolyan (Adult Blood Disorders), Yerevan
  - Hematology Center After Prof. R. Yeolyan (Clinic of Adults Oncology), Yerevan
  - National Center of Oncology Named After V.A. Fanarjyan, Yerevan
- Austria (2):
  - Wiener Gesundheitsverbund - Klinik Hietzing 06 FE Study, Vienna
  - Wiener Gesundheitsverbund - Klinik Hietzing 06 Study, Vienna
- Bulgaria (2):
  - Complex Oncology Center - Plovdiv - Base II, Plovdiv
  - Specialized Hospital for Active Treatment of Hematological Disease EAD, Sofia
- Canada (5):
  - University of Alberta Hospital, Edmonton
  - QEII Health Sciences Centre, Nova Scotia
  - The Ottawa Hosptial, Ottawa
  - Sunnybrook Health Sciences Centre, Toronto
  - Princess Margaret Cancer Center, Toronto
- Hôpital Emile Muller, Mulhouse, Grand Est, France
- Germany (2):
  - Städtisches Klinikum Braunschweig, Braunschweig, Lower Saxony
  - Universitätsklinikum Schleswig-Holstein - Campus Lübeck, Lübeck, Schleswig-Holstein
- Debreceni Egyetem Klinikai Kozpont, Belgyogyszati Klinika, B epulet, Hematologia, Debrecen, Hungary
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy
- Centrum Badań Klinicznych Piotr Napora Lekarze Sp. p., Wroclaw, Lower Silesian Voivodeship, Poland
- Romania (2):
  - Institutul Oncologic Bucuresti - Prof. Dr. Alexandru Trestioreanu, Bucharest
  - Institutul Oncologic Prof. Dr. Ion Chiricuta, Cluj-Napoca
- Summit Clinical Research s.r.o, Bratislava, Slovakia
- Spain (5):
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Clínica Universidad de Navarra - Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No